CLINICAL TRIAL: NCT01611324
Title: Efficacy of Alkalinised 2% Mepivacaine for Local Infiltration Anesthesia, in Ambulatory Phlebectomy
Brief Title: Painless Local Infiltration Anesthesia
Acronym: EASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Raffaele Antonelli Incalzi, Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EASE
Record Dates: First submitted 2012-05-17; First posted 2012-06-04 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Varicose Veins; Pain; Surgery; Anesthesia
Keywords: Varicose Veins; Phlebectomy; Local Anesthesia
MeSH Terms: conditions — Varicose Veins; Pain | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alkalinised anesthetic solution (Experimental)
  Interventions: Drug: Mepivacaine chlorhydrate 2% in Sodium Bicarbonate 1.4%
- Non alkalinised anesthetic solution (Active Comparator)
  Interventions: Drug: Mepivacaine chlorhydrate 2% with epinephrine in NS 0.9%

INTERVENTIONS:
Drug: Mepivacaine chlorhydrate 2% in Sodium Bicarbonate 1.4% — 4 mL mepivacaine chlorhydrate 20 mg/mL with epinephrine 5 mcg/mL diluted with 16 mL sodium bicarbonate 1.4%
  Other Names: Carbosen© 2%
  Arms: Alkalinised anesthetic solution
Drug: Mepivacaine chlorhydrate 2% with epinephrine in NS 0.9% — 4 mL mepivacaine chlorhydrate 20 mg/mL with epinephrine 5 mcg/mL diluted with 16 mL sodium chloride 0.9%
  Other Names: Carbosen© 2%
  Arms: Non alkalinised anesthetic solution

SUMMARY:
The purpose of this study is to assess if a dilution with 1.4% sodium bicarbonate of a 2% mepivacaine+epinephrine solution, can be effective in reducing the pain associated with local infiltration anesthesia, during ambulatory phlebectomy procedures.

DETAILED DESCRIPTION:
The use of local anesthesia by infiltration (LIA), usually prepared with 1% lidocaine or mepivacaine 2%, in combination with epinephrine and diluted with saline solution, it's commonly performed in ambulatory phlebectomy procedures.

Although this kind of anesthesia is among the most effective and safe available, the infiltration of local anesthetic is accompanied by pain in the majority of patients. This can be particularly important in ambulatory phlebectomy procedures, where large areas need to be anesthetized.

Numerous methods have been proposed to alleviate the pain associated with LIA, such as reducing the rate of administration or warming the anesthetic solution.

Sodium bicarbonate added in small concentrations, can also be effective in reducing significantly the pain associated with LIA. A recent trial has confirmed the viability and effectiveness of a solution of lidocaine 1% diluted in sodium bicarbonate 1.4%, in varicose vein surgery.

The purpose of this study is to evaluate the effectiveness in alleviating the pain associated with LIA, of a solution of mepivacaine 2%+epinephrine diluted with sodium bicarbonate 1.4%, compared with an analogous solution diluted with normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ambulatory phlebectomy

Exclusion Criteria:

* Allergy to amide anesthetics
* Sinoatrial node disease or any degree of atrio-ventricular block
* Acute diseases
* Chronic kidney or liver disease
* Treatment with drugs that alter pain sensitivity (e.g. analgesics)
* Treatment with monoamine oxidase inhibitors or tricyclic antidepressants
* Major psychiatric disorders according to DSM IV-TR diagnostic criteria
* Alcohol abuse actual or recent as described in DSM IV-TR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | Initial 2 minutes of the procedure
  Pain severity will be rated by the subjects on a visual analog scale, after the first five injections (placement of the needle + administration of anesthetic solution).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ricci, M.D., Study Chair — University Campus Bio-Medico; Leo Moro, M.D., Principal Investigator — University Campus Bio-Medico; Francesco Maria Serino, M.D., Principal Investigator — University Campus Bio-Medico; Raffaele Antonelli Incalzi, M.D., Study Director — University Campus Bio-Medico
Locations (1):
- Policlinico Universitario Campus Bio-Medico, Rome, RM, Italy

REFERENCES:
- [Background] Creton D, Rea B, Pittaluga P, Chastanet S, Allaert FA. Evaluation of the pain in varicose vein surgery under tumescent local anaesthesia using sodium bicarbonate as excipient without any intravenous sedation. Phlebology. 2012 Oct;27(7):368-73. doi: 10.1258/phleb.2011.011026. Epub 2011 Nov 21. PMID 22106448